CLINICAL TRIAL: NCT05310903
Title: A Multi-Centre Survey on Hospital Malnutrition in Afghanistan
Brief Title: Prevalence of Hospital Malnutrition in Afghanistan
Acronym: ANSH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kateb University (Other)
Collaborators: Afghanistan Medical Council (Unknown)
Responsible Party: Principal Investigator, Jaffer Shah, Principle Investigator, Clinical Researcher, Medical Research Center, Kateb University
Other Study IDs: 51231301
Record Dates: First submitted 2022-03-14; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Malnutrition
Keywords: Malnutrition; Nutrition Disorders
MeSH Terms: conditions — Malnutrition; Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the prevalence of malnutrition among adult patients in hospitals across Afghanistan.

DETAILED DESCRIPTION:
Malnutrition is associated with negative patient outcomes and increased healthcare costs. The purpose of this cross-sectional study is to determine the prevalence of malnutrition at admission or discharge in adult patients in hospitals across Afghanistan. The secondary outcome is to assess risk factors for malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* All admitted or discharged patients age 18-65
* Males and females
* Conscious
* Informed consent provided

Exclusion Criteria:

* Patients undergoing surgery on the data collection day
* Outpatients
* Pregnant females
* Pediatric patients Patients with psychiatric or eating disorders Patients on dialysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted or discharged from hospitals in Afghanistan during the defined study period will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Malnutrition | Baseline
  Nutrition status will be measured with the subjective global assessment (SGA).The SGA tool categorizes nutritional status as: well-nourished (SGA-A), moderately malnourished (SGA-B), and severely malnourished (SGA-C).

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Shah, Principal Investigator — Medical Research Center, Kateb University

IPD SHARING:
Plan to Share IPD: Undecided